CLINICAL TRIAL: NCT00002368
Title: An International, Double Blind, Randomized, Phase III Study to Evaluate the Tolerance, Safety, and Effectiveness of Viramune (Nevirapine) in Preventing Clinical AIDS Progression Events or Death When Used in Combination With Lamivudine (3TC) and Stable (>= 4 Weeks) Background Nucleoside Therapy
Brief Title: The Safety and Effectiveness of Nevirapine Plus Lamivudine Plus Other Anti-HIV Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 200E; 1100.1090
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Nevirapine; Lamivudine; Disease Progression; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Disease Progression | interventions — Nevirapine; Lamivudine

INTERVENTIONS:
Drug: Nevirapine
Drug: Lamivudine

SUMMARY:
To evaluate the tolerance, safety, and effectiveness of Viramune in preventing clinical AIDS progression events or death when used in combination with Lamivudine and background nucleoside therapy.

DETAILED DESCRIPTION:
Eligible patients will be randomized to treatment with either 1) open-label 3TC twice daily plus Viramune once daily for 2 weeks and then with Viramune twice daily; or 2) open label 3TC twice daily plus Viramune placebo once daily for 2 weeks and then twice daily Viramune. Patients will start Viramune and 3TC on study day 0. Patients will be evaluated for development of AIDS progression events at months 1, 2, 3, and 4, and every 2 months thereafter until 18 months after the last patient is enrolled or 24 months, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4+ cell count <= 200 cells/mm3.
* Life expectancy > 3 months.
* Written informed consent from parent or guardian for patients < 18 years of age.
* Willingness and ability to follow protocol requirements.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following conditions or symptoms are excluded:

Patient is enrolled or plans to enroll during the course of this study in another clinical study of an antiretroviral or other agent used to treat HIV-1 infection.

* NOTE:
* Patients are allowed to participate in opportunistic infection clinical studies if the investigational agent is not contraindicated for the study.

Concurrent Medication:

Excluded:

* Patient is receiving therapy with an antiretroviral agent other than ZDV, d4T, ddI, ddC, or 3TC.
* Patient is receiving acute therapy for a clinical AIDS progression event such as systemic chemotherapy.
* Dicumarol, Warfarin and other anticoagulant medications.
* Tolbutamide.
* Investigational drugs (unless included in opportunistic infection clinical trial) and all antiretroviral agents (excluding ZDV, ddC, ddI, d4T and 3TC).
* Neurotoxic drugs.
* Cimetidine.
* Erythromycin.

Concurrent Treatment:

Excluded:

Radiation therapy.

Patients with any of the following prior conditions and symptoms are excluded:

History of clinically important disease other than HIV-1 infection or related diseases that, in the opinion of the investigator, may put the patient at risk because of participation in this study.

Prior Medication:

Excluded:

* Patient has received prior therapy with Viramune or any other non-nucleoside reverse transcriptase inhibitor.
* Patient has received any immunosuppressive or cytotoxic drugs or any other experimental agent within 4 weeks prior to study day 1.
* Patient has received treatment with erythromycin, coumadin/warfarin, phenobarbital, amoxicillin/clavulanic acid, or ticarcillin/clavulanic acid within 2 weeks prior to study day 0.

Risk Behavior:

Excluded:

Patients who are active chronic alcohol or substance abusers or have an active psychiatric condition sufficient to impair compliance with protocol requirements.

Required:

Patient must be receiving stable nucleoside therapy with at least one agent for >= 4 weeks prior to study day 0. Zidovudine (ZDV), Zidovudine + Dideoxycytidine (ddC), or Zidovudine + Didanosine (ddI) must be used unless prior intolerance precludes ZDV use. Stable use means no change in dose > 50% for any background nucleoside within four weeks prior to study day 0.

NOTE:

* If patient is ZDV intolerant, ddC, ddI or D4T monotherapy is allowed.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000

CONTACTS AND LOCATIONS:
Locations (53):
- United States (53):
  - Drug Research and Analysis Corp, Montgomery, Alabama
  - Dr G Michael Wool, Los Angeles, California
  - UCLA School of Medicine / Ctr for Research and Education, Los Angeles, California
  - AIDS Research Ctr / Palo Alto VA Health Care System, Palo Alto, California
  - AIDS Community Research Consortium, Redwood City, California
  - ViRx Inc, San Francisco, California
  - San Francisco Gen Hosp / UCSF AIDS Program, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Infectious Disease Specialists, Colorado Springs, Colorado
  - Denver Public Health, Denver, Colorado
  - Dr Miguel Mogyoros / Clinical Research Dept, Denver, Colorado
  - Wilmington Hosp, Wilmington, Delaware
  - Novum Inc, Washington D.C., District of Columbia
  - Anthony LaMarca, Fort Lauderdale, Florida
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Dr Robert Schwartz, Fort Myers, Florida
  - McGregor Clinic / Lee County Public Health Unit, Fort Myers, Florida
  - P Andrew Coley, Jacksonville, Florida
  - Goodgame Med Group, Maitland, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Palm Beach Research Ctr, West Palm Beach, Florida
  - Dr John Pottage, Chicago, Illinois
  - Northwestern Univ / Division of Infectious Diseases, Chicago, Illinois
  - Rush Presbyterian / Saint Luke's Med Ctr / Infect Dis, Chicago, Illinois
  - Indiana Univ Med School, Indianapolis, Indiana
  - Dr Daniel H Gervich, Des Moines, Iowa
  - Univ of Iowa, Iowa City, Iowa
  - Univ of Kentucky Med Cntr / Dept of Med / Div of ID, Lexington, Kentucky
  - Med Research Ctr, New Orleans, Louisiana
  - New England Med Ctr, Boston, Massachusetts
  - Beth Israel Hosp / Virology Research Clinic, Boston, Massachusetts
  - New England Deaconess Hosp, Boston, Massachusetts
  - International Medicine and Infectious Disease, Minneapolis, Minnesota
  - Trinity Lutheran Hosp / HIV Program, Kansas City, Missouri
  - Infectious Disease Associates of Central New Jersey, Somerville, New Jersey
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Dr David Kaufman, New York, New York
  - Saint Vincent Med Ctr, Staten Island, New York
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - The Research and Education Group, Portland, Oregon
  - Hershey Med Ctr / Dept of Med / Div of Hematology, Hershey, Pennsylvania
  - Univ of Pennsylvania / Division of Infectious Diseases, Philadelphia, Pennsylvania
  - Novum Inc, Pittsburgh, Pennsylvania
  - Omega Med Research, Providence, Rhode Island
  - Med Univ of South Carolina / Div of Infect Dis, Charleston, South Carolina
  - Dr Alfred Burnside, Columbia, South Carolina
  - Dr Susie Sargent, Memphis, Tennessee
  - Nelson Tebedo Health Resource Ctr, Dallas, Texas
  - Univ of Texas Med Branch / Div of Infectious Dis, Galveston, Texas
  - Houston Clinical Research Network / Div of Montrose Clinic, Houston, Texas
  - Walter Gaman, Irving, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Advanced Research Management, Seattle, Washington